CLINICAL TRIAL: NCT04903106
Title: A Prospective, Multi-center Clinical Study to Evaluate the Safety and Performance of the FAST-FIX FLEX System for Meniscal Repairs (MR) and Meniscal Allograft Transplantations (MAT)
Brief Title: Safety and Performance Study of the FAST-FIX FLEX System for Meniscal Repairs and Meniscal Transplantations
Acronym: FAST-FIX FLEX
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: FAST-FIX FLEX.2020.09
Record Dates: First submitted 2021-05-19; First posted 2021-05-26 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Meniscus Tear
Keywords: FAST-FIX FLEX; meniscal; meniscus; knee repair; meniscal allograft transplant; all-inside meniscal repair; FASTFIX

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Meniscal Tear: Subject requires a meniscus repair concerning the red-red or red-white zones for acute or chronic 1-, 2- or 3-segment lesions, with or without associated anterior cruciate ligament (ACL) reconstruction.
  Interventions: Device: FAST-FIX FLEX Meniscal Repair System
- Meniscal Insufficiency: Subject requires a MAT for symptomatic meniscal insufficiency (load related pain and swelling in the compartment undergoing meniscectomy) for which conservative treatment has failed.
  Interventions: Device: FAST-FIX FLEX Meniscal Repair System

INTERVENTIONS:
Device: FAST-FIX FLEX Meniscal Repair System — Standard of care surgery in which the meniscus is repaired using FAST-FIX FLEX device.
  Groups: Meniscal Tear
Device: FAST-FIX FLEX Meniscal Repair System — Standard of care surgery in which the FASTFIX FLEX device is used during the meniscal allograft transplantation procedure.
  Groups: Meniscal Insufficiency

SUMMARY:
This study is a post-market follow-up study (PMCF). The data collected will serve the purpose of confirming the safety and performance of the FAST-FIX FLEX device, used according to the indicated for use (IFU) for meniscal repair and meniscal transplantations. Data will be collected on patients prior to surgery, at surgery and for 12 months after surgery.

DETAILED DESCRIPTION:
This PMCF study is to satisfy the post-market surveillance obligations to the European Medical Device Regulation (EU MDR 2017/745). The data collected will serve the purpose of confirming the safety and performance of the FAST-FIX FLEX device, used according to the indicated for use (IFU) for meniscal repair and meniscal transplantations. Data will be collected on patients prior to surgery, at surgery and for 12 months after surgery.

The objectives of the study are to assess the clinical success rate of both clinical indications (meniscal repair and meniscal allograft transplantations) and the performance and safety of the FAST-FIX FLEX meniscal repair system.

The sample size for this study is precision-based and not based on statistical power considerations. Thus, no formal statistical hypothesis is formulated. The sample size for this study is determined based on the feasibility of recruitment, enrolment and follow-up considerations.

The primary endpoint upon which the sample size is determined is defined by the rate of reoperation after at 12 months.

Additionally, secondary endpoints in this study assess success rate, meniscus healing and clinical performance of Patient Reported Outcomes (PRO) for meniscal repair and meniscal allograft transplantations.

ELIGIBILITY:
Meniscal Repair Inclusion Criteria:

1. Subject provides written informed consent for study participation using an independent ethical committee (IEC) / institutional review board (IRB) approved consent form;
2. Subject is between sixteen (16) and seventy (70) years of age, inclusive at the time of screening;
3. Subject is willing and able to participate in required follow-up visits and is able to complete study activities;
4. Subject requires a meniscal repair;
5. Subject is suitable to participate in the study in the opinion of the Investigator;
6. Subject requires a meniscus repair concerning the red-red or red-white zones for acute or chronic 1-, 2- or 3-segment lesions, with or without associated anterior cruciate ligament (ACL) reconstruction.

Meniscal Allograft Transplantation Inclusion Criteria:

1. Subject provides written informed consent for study participation using an independent ethical committee (IEC) / institutional review board (IRB) approved consent form;
2. Subject is between sixteen (16) and seventy (70) years of age, inclusive at the time of screening;
3. Subject is willing and able to participate in required follow-up visits and is able to complete study activities;
4. Subject requires a meniscal allograft transplantation;
5. Subject is suitable to participate in the study in the opinion of the Investigator.
6. Subject requires a MAT for symptomatic meniscal insufficiency (load-related pain and swelling in the compartment post meniscectomy) for which conservative treatment has failed, with or without cartilage repair or restoration (including ACL reconstruction or repair).

Meniscal Repair Exclusion Criteria:

1. Contraindications (per the FAST-FIX FLEX IFU) or hypersensitivity to the use of the FAST-FIX FLEX implant material. Where material sensitivity is suspected, appropriate tests should be made and sensitivity ruled out prior to implantation;
2. Enrolled in the treatment period of another clinical trial within thirty (30) days of operative visit, or during the study;
3. Women who are pregnant or nursing;
4. Any subject that meets the definition of a Vulnerable Subject per ISO 14155 Section 3.55 (except for subjects aged sixteen (16) or seventeen (17) years of age with consent from their legally authorized representative);
5. Subjects with a history of poor compliance with medical treatment, physical therapy (PT)/rehabilitation, or clinical study participation;
6. Patients with irreparable meniscal tears (i.e. multiple tears);
7. Subjects with full thickness cartilage defects greater than 10mm in diameter and/or serious defects;
8. Patients with concomitant ligament injuries that do not require surgical repair (i.e. ACL with Grade 3 lateral collateral ligament (LCL) injury or medial collateral ligament (MCL) injury);
9. Performance of a significant concomitant procedure, specifically a cartilage repair or restoration (excluding ACL reconstruction or repair, lateral extra-articular tenodesis, anterolateral ligament (ALL) reconstruction) intended as a therapeutic intervention on the study knee;
10. History of ipsilateral knee surgery, septic joint, or fracture;
11. Pathological conditions in the soft tissue that would prevent secure fixation of the device;
12. Physical conditions which would eliminate, or tend to eliminate, adequate anchor support or retard healing;
13. The presence of infection;
14. Conditions which would limit the patient's ability or willingness to restrict activities or follow directions during the healing period;
15. Malalignment: genu varus and genu valgus angles greater than 5° as evaluated by the patient's physician as per their standard of care;
16. Patients who have an Ahlback grade greater than II;
17. Patients with a body mass index larger than 35;
18. Subjects with a medical or physical condition that, in the opinion of the Investigator, would preclude safe subject participation in the study.

Meniscal Allograft Transplantation Exclusion Criteria:

1. Contraindications (per the FAST-FIX FLEX IFU) or hypersensitivity to the use of the FAST-FIX FLEX implant material. Where material sensitivity is suspected, appropriate tests should be made and sensitivity ruled out prior to implantation;
2. Enrolled in the treatment period of another clinical trial within thirty (30) days of operative visit, or during the study;
3. Women who are pregnant or nursing;
4. Any subject that meets the definition of a Vulnerable Subject per ISO 14155 Section 3.55 (except for subjects aged sixteen (16) or seventeen (17) years of age with consent from their legally authorized representative);
5. Subjects with a history of poor compliance with medical treatment, physical therapy (PT)/rehabilitation, or clinical study participation;
6. Patients with concomitant ligament injuries that do not require surgical repair (i.e. ACL with Grade 3 lateral collateral ligament (LCL) injury or medial collateral ligament (MCL) injury);
7. Performance of a significant concomitant procedure (excluding ACL reconstruction or repair, lateral extra-articular tenodesis, anterolateral ligament (ALL) reconstruction) intended as a therapeutic intervention on the study knee;
8. History of ipsilateral knee surgery, septic joint, or fracture (excluding MAT indication);
9. Pathological conditions in the soft tissue that would prevent secure fixation of the device;
10. Physical conditions which would eliminate, or tend to eliminate, adequate anchor support or retard healing;
11. The presence of infection;
12. Conditions which would limit the patient's ability or willingness to restrict activities or follow directions during the healing period;
13. Malalignment: genu varus and genu valgus angles greater than 5° as evaluated by the patient's physician as per their standard of care;
14. Patients who have an Ahlback grade greater than II;
15. Patients with a body mass index larger than 35;
16. Subjects with a medical or physical condition that, in the opinion of the Investigator, would preclude safe subject participation in the study.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who require a meniscal repair or meniscal allograft transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2024-11-26 (Actual)

PRIMARY OUTCOMES:
Clinical Success | 12 months
  Rate of reoperation due to meniscal repair failure at 12 months postoperative

SECONDARY OUTCOMES:
Clinical Success | 6 months
  Rate of reoperation due to meniscal repair failure at 6 months postoperative
Clinical Success | 6 months and 12 months
  Rate of reoperation due to meniscal allograft transplantation failure at 6 months & 12 months post-operative
Meniscal Healing | Pre-operatively, 6 months and 12 months
  MRI to assess structural integrity and meniscal healing at 6 months and 12 months
Change in Patient Reported Outcome (PRO): International Knee Documentation Committee (IKDC) Subjective Score | Pre-operatively, 6 months and 12 months
  The International Knee Documentation Committee (IKDC) Subjective score was developed to detect improvement or deterioration in symptoms, function, and sports activities due to knee impairment, including patients with meniscal injuries. There are three domains:
  1. symptoms, including pain, stiffness, swelling, locking/catching, and giving way (7 items),
  2. sports and daily activities (10 items), and
  3. current knee function and knee function prior to knee injury (1 item, not included in the score).
  Responses vary for each item. The possible score ranges from 0-100,where 100 = no limitation with daily or sporting activities and the absence of symptoms.
Change in Patient Reported Outcome (PRO): Lysholm Score | Pre-operatively, 6 months and 12 months
  This tool measures the domains of symptoms and complaints and functioning of daily activities. The scale consists of 8 items and is scaled from 0 to 100, with a higher score indicating fewer symptoms and higher level of functioning.
Change in Patient Reported Outcome (PRO): EuroQol 5 Dimension 5 Level (EQ-5D-5L) | Pre-operatively, 6 months and 12 months
  The EQ-5D-5L descriptive system comprises the following dimensions: Mobility, Self-Care, Usual Pain/ Discomfort and Anxiety/ Depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems.

CONTACTS AND LOCATIONS:
Overall Officials: Rupali Soeters, Study Chair — Smith & Nephew, Inc.
Locations (5):
- United States (2):
  - Rush University Medical Center, Chicago, Illinois
  - Hospital for Special Surgery, New York, New York
- Fremantle Hospital, Fremantle, Western Australia, Australia
- Ambroise Paré Clinic, Paris, Neuilly-Sur-Seine, France
- Robert Jones and Agnes Hunt Orthopaedic Hospital NHS Foundation Trust, Oswestry, Shropshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No